CLINICAL TRIAL: NCT03985592
Title: ICU BEREAVE: Feasibility of a Multi-component Bereavement Support Intervention to Prevent Severe Grief Reaction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The investigators experienced several barriers: including COVID-19 delays on research, high staff turnover, and burnout amongst ICU Nursing Staff. The study team and ICU staff determined low feasibility of completing Phase 2, 3, and 4 as a result.
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Virtual Hospice (Unknown)
Responsible Party: Principal Investigator, James Downar, Head of the Division of Palliative Care, Ottawa Hospital Research Institute
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 1466
Record Dates: First submitted 2019-06-07; First posted 2019-06-13 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Severe Grief Reaction
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: The multi-component intervention aims to evaluate the feasibility as well as success of imparting educational knowledge and applied techniques to ICU clinicians (i.e., physicians, RNs, social workers) on how to support bereaved FMs. The overall purpose of the intervention is to optimize preemptive strategies in reducing SGRs in FMs. To determine the effectiveness of this intervention a series of standardized and validated measures of wellbeing will be given to FMs after the typical bereavement period ends. The intervention is designed to be implementable in any ICU setting across Canada and potentially abroad.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Educational Intervention for ICU-Based Clinicians (Other): ICU-based clinicians (e.g. physicians, RNs, and social workers) will be provided with educational modules related to bereavement support for family members. Following the modules a survey will be provided to participants to assess their perceived usefulness of the modules.
  Interventions: Behavioral: Education
- Educational material and personalized card of condolence (Experimental): Members of the ICU team who cared for deceased ICU patients will be asked to send a letter of condolence to family members listed as the patient's primary contact and provide them with educational modules related to bereavement support for family members.
  Interventions: Behavioral: Education
- Virtual meeting with the care team to address unmet needs (Experimental): At 8-12 weeks post-death, the study team will contact FMs and invite them to meet virtually with the care team. Our observational studies indicated that the most common need reported by bereaved FMs was the desire to meet with the care team to review events during the ICU stay and particularly the events that led to death, and that this was the type of support that ICU clinicians were most comfortable providing.
  Interventions: Behavioral: Education
- Offering a facilitated storytelling intervention session (Experimental): At six months post-death, the study team will contact FMs and administer the Inventory of Complicated Grief-Revised (ICG-r), Brief Grief Questionnaire (BGQ), Impact of Events Scale - Revised (IES-r), Patient Health Questionnaire-9 (PHQ-9), and the Bereavement Dependency Scale (BDS). FMs who complete all questionnaires will be invited to participate in a 1-2-hour narrative exploration of their grief and bereavement experience, regardless of the severity of their symptoms. Those with severe symptoms will be notified of symptom severity, and offered to participate in the narrative exploration of their grief and bereavement experience. Storytelling interventions require specialized resources but the results of Barnato et al., as well as the response to our qualitative interviews, suggest that this intervention may only be helpful for selected FMs. Storytelling interventions have been shown to reduce healthcare utilization and improve subjective health following a traumatic experience.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education — Intervention description provided in elaboration on arms of the study.
  Other Names: Bereavement support, social, and SGR risk assessment

SUMMARY:
Nearly 1% of the Canadian population dies every year. When people die, their bereaved family members (FMs) normally experience grief that diminishes over time and without serious psychological or medical impairment. However, some FMs experience a severe grief reaction (SGR) with intense symptoms and impairment lasting months or years; this is more common among FMs of those who die in the Intensive Care Unit (ICU). Many bereaved FMs would like to have bereavement support, and many ICU organizations identify bereavement support as a clinical and research priority, yet few ICUs provide routine support.

In order to determine the feasibility and acceptability of a complex support intervention for bereaved FMs, the investigators will pilot a multi-component bereavement intervention through a mixed-methods study. Methods will include a series of semi-structured interviews, questionnaires and narrative therapy sessions. The target population for this study is both ICU clinical staff (e.g. physicians, registered nurses [RN], allied health professionals) and FMs of relatives who died in the ICU. The intervention is premised on a robust series of educational modules aimed at increasing ICU staff members' knowledge of and level of comfort with bereavement support ICU FMs.

In a previous study, the investigators have established that SGRs can be predicted using screening tools early after the loss, and that ICU-based clinicians are eager to provide bereavement support. There are effective treatments for SGRs once they have been diagnosed after 6 months, but this can mean many months of suffering for the FM. In this project, the investigators plan to develop and test the feasibility of an early bereavement support program that follows bereaved FMs after a loss, provides information and support, and uses effective therapies aimed at preventing the development of a SGR.

DETAILED DESCRIPTION:
Almost 1% of the population dies annually. When people die, it is normal for their bereaved family members (FMs) to experience grief. This grief usually diminishes, but in some cases FMs suffer from severe grief reaction (SGR) with intense yearning or separation distress, as well as emotional, cognitive and functional impairment lasting months or years. SGRs are linked with declining health, increased use of healthcare resources, and even death. ICU deaths are associated with a higher incidence of SGR2 - symptoms of psychiatric illness and have been reported in 34-67% of surviving FMs with 22% experiencing significant social distress.

As grieving death is an expected human response, SGRs cannot be diagnosed until >6 months after a loss, but the investigators found that a SGR at 6 months can be accurately predicted by screening tests 3 months after a death. Early identification provides opportunity for early intervention with the hope of preventing or reducing the severity of SGRs. There are effective treatments for established SGRs (i.e. >6 months post-death), including psychotherapy tailored to SGR. This therapy works through 3 mechanisms: (1) by encouraging exposure to reminders and situations that the FM is avoiding, (2) restructuring through reconstructing an understanding of the loss and grief experience, and (3) behavioural activation to re-establish social interaction. Some ICU-based support interventions administered pre-death are effective in reducing psychological morbidity, while others have shown no effect or even harm.

Many bereaved FMs would appreciate bereavement support, and ICU organizations have identified bereavement support as a clinical and research priority. Yet few ICUs have devoted resources toward bereavement screening or support. Our previous multi-centre study found that only 16% of Canadian ICU clinicians follow up with FMs after a death, and bereaved FMs rarely, if ever, report being contacted after the death of their loved one. Few ICU clinicians have received formal training in bereavement support and many report "not knowing what to say" in response to strong emotions.

Currently, less than half of Canadian ICU clinicians (physicians and registered nurses [RN]) are comfortable providing any form of bereavement support to FMs at the time of death, and fewer than 18% perceive that FMs may have social or informational needs following a death. Similarly, FMs are often unwilling or unable to access bereavement support even when resources are available with over half of eligible participants declining participation in ICU-based bereavement interventions.

Single interventions are not effective for preventing SGRs in unselected populations of bereaved FMs (thought may benefit high-risk populations). Thus our pilot project will combine several promising scalable and low-resource interventions in a "bundle", to improve the chances of meeting these needs and overcoming these barriers. As a research-based intervention, this study will examine the feasibility of implementing measures to reduce SGRs while also determining the best methods to address the social and educational needs of clinicians and FM.

ELIGIBILITY:
Inclusion Criteria:

* A family member of a recently deceased patient at the Ottawa Hospital ICU

Exclusion Criteria:

* Non-Family Member
* Death not in ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-02-02 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-02-07 (Actual)

PRIMARY OUTCOMES:
The Inventory of Complicated Grief-Revised (ICG-r) | At 6 months post death
  Indicates rate of pathological grief. A total of 19 questions. Respondents rate the frequency with which they experience each item on a 5-point scale (0-4), ranging from "never" to "always." Respondents with ICG scores greater than 25 are significantly more impaired in social, general, mental and physical health functioning and in bodily pain than those with ICG scores less than or equal to 25. Higher scores result in higher likelihood of CG.
Brief Grief Questionnaire (BGQ) | At 6 months post death
  A self reporting instrument assessing complicated grief. A total of 5 questions on a 3 point scale. A total score of 10 is possible. Higher scores result in higher likelihood of CG.
Impact of Events Scale - Revised (IES-r) | At 6 months post death
  A self reporting instrument that assesses subjective distress caused by traumatic events. Items are rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). The IES-R yields a total score (ranging from 0 to 88) and subscale scores can also be calculated for the Intrusion, Avoidance, and Hyperarousal subscales. Higher scores are linked with a greater likelihood of distress
Patient Health Questionnaire-9 (PHQ-9) | At 6 months post death
  A multipurpose instrument for screening for severity of depression. A total of 9 questions. Respondents answer from "0" to "4" for each question. The total range is from 0 to 36. A higher score is correlated with greater level of depression.
Bereavement Dependency Scale (BDS) | At 6 months post death
  Used as a predictor of enduring and complicated grief. A total of 6 questions. Items are rated on a 5 point scale from "1" to "5". A higher score is linked to dependency on deceased.

CONTACTS AND LOCATIONS:
Overall Officials: James Downar, MD, Principal Investigator — Physician; Brandi Vanderspank-Wright, Phd,RN, Principal Investigator — Investigator
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
All participant data will be kept securely by the research team and de-identified for any future publication.